CLINICAL TRIAL: NCT03390127
Title: Effect of Positive End-expiratory Pressure on Arterial Oxygen Partial Pressure in Elderly Patients Undergoing Urologic Surgery Using LMA Supreme™ in Lithotomy Position
Brief Title: Effect of PEEP on Arterial Oxygen Partial Pressure in Elderly Patients With Lithotomy Position Using LMA Supreme™
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Asan Medical Center (Other)
Responsible Party: Principal Investigator, Young-Kug Kim, Professor, Asan Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: 2017-1397
Record Dates: First submitted 2017-12-26; First posted 2018-01-04 (Actual); Last update posted 2018-04-06 (Actual); Status verified 2018-04

CONDITIONS: Urinary Bladder Neoplasms; Prostatic Neoplasms
Keywords: elderly; lithotomy position; PEEP; laryngeal mask airway
MeSH Terms: conditions — Urinary Bladder Neoplasms; Prostatic Neoplasms

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group P (Experimental): After LMA Supreme™ insertion, PEEP of 7 cmH2O would apply during general anesthesia with mechanical ventilation.
  Interventions: Other: PEEP
- Group Z (No Intervention): After LMA Supreme™ insertion, PEEP would not apply during general anesthesia with mechanical ventilation.

INTERVENTIONS:
Other: PEEP — After LMA Supreme™ insertion, it's proper position is confirmed. Then, PEEP of 7 cmH2O is applied during mechanical ventilation.
  Other Names: Application of PEEP 7 cmH2O
  Arms: Group P

SUMMARY:
The purpose of the present study is to compare the effect of PEEP on arterial oxygen partial pressure in elderly patients undergoing urologic surgery using LMA supreme™ in a lithotomy position.

DETAILED DESCRIPTION:
Positive end-expiratory pressure (PEEP) during general anesthesia with mechanical ventilation is routinely used as a standard lung protective strategy to prevent postoperative pulmonary complications including atelectasis.

In urologic surgery, elderly patients are common. Since aging decreases the elasticity of lung tissues and allowing the collapse of small airways, old age is a risk factor for postoperative atelectasis. Lithotomy position is the preferred position in urologic surgery. However, it causes the abdominal viscera to displace the diaphragm cephalad, reducing lung compliance and resulting atelectasis. Therefore, in elderly patients undergoing urologic surgery with lithotomy position, PEEP may be essential to prevent postoperative atelectasis.

Laryngeal mask airway (LMA) has been widely used in urologic surgery with lithotomy position because of short surgical time and no necessity of administration of muscle relaxant. However, application of PEEP when using LMA is still controversy. Therefore, in the present study, we aimed to compare the effect of PEEP on arterial oxygen partial pressure in elderly patients undergoing urologic surgery using LMA supreme™ in a lithotomy position.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing urologic surgery with lithotomy position under general anesthesia
* Elderly patients (65 ≤ Age < 80)
* American Society of Anesthesiologists (ASA) physical status: 1-3
* Patients who voluntarily agreed to participate in this clinical study

Exclusion Criteria:

* Heart failure (ejection fraction ≤ 40%)
* Hemodynamic instability during perioperative period
* Lung diseases (chronic obstructive pulmonary disease, asthma, bullae, pleural effusion)
* Obesity (BMI ≥ 30 kg/m2)
* Neck or upper respiratory tract pathologies
* An increased risk of pulmonary aspiration
* Anticipation of the difficult laryngeal mask fixation due to poor dentition

Ages: 65 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 68 (Actual)
Dates: Start 2018-01-05 (Actual); Primary Completion 2018-03-14 (Actual); Study Completion 2018-03-21 (Actual)

PRIMARY OUTCOMES:
The difference of arterial oxygen partial pressure (PaO2) between group P and group Z | 1 hour after LMA insertion
  The difference of arterial oxygen partial pressure (PaO2) between group P and group Z 1 hour after LMA insertion by arterial blood gas analysis

SECONDARY OUTCOMES:
Postoperative pulmonary complications | Up to seven days
  Postoperative pulmonary complications include atelectasis, pneumothorax, bronchospasm, pneumonia, pulmonary edema, pleural effusion, respiratory failure
Complications associated with LMA | 1 hour after end of surgery
  Complications associated with LMA include oropharyngolaryngeal injury and sore throat.
Incidence of significant leak of LMA | At 5, 30, 60 mins after LMA insertion
  Significant leak of LMA means that leak friction is more than 0.2.

CONTACTS AND LOCATIONS:
Overall Officials: Young-Kug Kim, MD, PhD, Principal Investigator — Asan Medical Center
Locations (1):
- Asan medical center, Seoul, South Korea